CLINICAL TRIAL: NCT05265117
Title: The Efficacy of Hyperthermic Intraperitoneal Chemotherapy to Ovarian Cancer Patients With Homologous Recombination Repair Defect and Residual: a Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-KY-073
Record Dates: First submitted 2022-03-02; First posted 2022-03-03 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2022-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIPEC: HIPEC is given after primary debulking surgery or interval debulking.
  Interventions: Procedure: HIPEC
- CONTROL: No HIPEC

INTERVENTIONS:
Procedure: HIPEC — HIPEC is given after primary or interval debulking surgery.
  Groups: HIPEC

SUMMARY:
Ovarian cancer is associated with the highest mortality of all gynecologic cancers. In patients with newly diagnosed advanced ovarian cancer after platinum-containing chemotherapy plus bevacizumab therapy, maintenance therapy with olaparib plus bevacizumab significantly prolongs progression-free survival (PFS) in the intended population and is recommended by guidelines. However, study shows those homologous recombinant repair defect (HRD) but Breast Cancer Susceptibility Gene(BRCA) wild type have limited benefit from maintenance therapy with olaparib plus bevacizumab when surgery is with residual(no-R0).

Can hyperthermic intraperitoneal chemotherapy(HIPEC) improve the benefits of first-line maintenance therapy in patients with non-R0 resection, HRD? The cohort study will enroll 310 patients with HRD and no-R0 resection who conduct HIPEC during primary treatment and then have olaparib plus bevacizumab as maintenance. Follow-up period is 30 months. The primary endpoint is PFS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Eastern Cooperative Oncology Group (ECOG) score 0-1
* Adequate kidney function (blood creatinine 58-96µmol/L)
* Adequate haematological function (haemoglobin ≥110g/L, leucocytes ≥4.0×109/L, neutrophils ≥2.0×109/L, platelets≥100×109/L)
* Adequate liver function (serum total bilirubin 3.4-22.2µmol/L, alanine aminotransferase (ALT) 7-40U/L, aspartate aminotransferase (AST) 13-35U/L, AST/ALT ≤1.5
* surgery with residual
* eligible to the maintenance therapy of olaparib plus bevacizumab

Exclusion Criteria:

* Expected life span ≤8 weeks
* Complicated with any other known malignancies
* Patients with dysfunction of swallow and digestion
* Patients who had received any kind of poly adenosinediphosphate-ribose polymerase（PARP）inhibitor
* refractory hypertension

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: high-grade serous ovarian cancer, International Federation of Gynecology and Obstetrics stage III-IV,HRD but BRCA wild type, chemotherapy regimen contains platinum and bevacizumab and then olaparib plus bevacizumab will be given as the maintenance therapy.
Sampling Method: Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
PFS | from the date of recruitment to the time of recurrence, assessed up to 30 months

SECONDARY OUTCOMES:
overall survival | from the date of recruitment to the time of death from any cause, assessed up to 30 months
adverse effect | from the date of recruitment up to 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No